CLINICAL TRIAL: NCT01100528
Title: Adjuvant Therapy for Patients With Primary Uveal Melanoma With Genetic Imbalance
Brief Title: Dacarbazine and Recombinant Interferon Alfa-2b in Treating Patients With Primary Uveal Melanoma With Genetic Imbalance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2609; NCI-2010-00640 (Other: NCI/CTRP)
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Ciliary Body and Choroid Melanoma, Medium/Large Size; Ciliary Body and Choroid Melanoma, Small Size; Iris Melanoma; Recurrent Intraocular Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Introns; Interferon alpha-2; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm I (Experimental): Patients receive dacarbazine IV on days 1 and 29. Beginning 4 weeks after the second dose of dacarbazine, patients receive recombinant interferon alfa-2b subcutaneously 3 times a week for 24 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: recombinant interferon alfa-2b; Drug: dacarbazine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: recombinant interferon alfa-2b — Given subcutaneously (SC) 3 times a week for 24 weeks
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; interferon alfa-2B; Intron A
Drug: dacarbazine — Given IV on days 1 and 29
  Other Names: Asercit; Biocarbazine; Dacarbazina Almirall; DIC; DTIC; DTIC-Dome
Other: laboratory biomarker analysis — Correlative studies obtained prior to therapy, every 8 weeks while on therapy, and then every 6 months during follow-up

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as dacarbazine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Recombinant interferon alfa-2b may interfere with the growth of tumor cells. Giving interferon alfa-2b together with dacarbazine may be an effective treatment for primary uveal melanoma.

PURPOSE: This phase II trial is studying how well giving dacarbazine together with recombinant interferon alfa-2b works in treating patients with primary uveal melanoma with genetic imbalance.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess disease-free survival (DFS) with sequential dacarbazine and interferon-alfa-2b as an adjuvant to primary therapy for patients with uveal melanoma with genetic imbalance.

SECONDARY OBJECTIVES:

I. Evaluate side effects and assess safety in the patient population.

II. Examine the relationship between the levels of plasma biomarkers of immune function and tumor invasion and the clinical outcome.

OUTLINE: Patients receive dacarbazine IV on days 1 and 29. Beginning 4 weeks after the second dose of dacarbazine, patients receive recombinant interferon alfa-2b subcutaneously 3 times a week for 24 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months.

ELIGIBILITY:
Inclusion

* Patients must have a diagnosis, either cytologic or histologic, of melanoma of the iris, ciliary body and/or choroid
* Patient's tumor must exhibit monosomy 3 and/or 8q amplification as determined by karyotype, comparative genomic hybridization (CGH), polymerase chain reaction (PCR)-based microsatellite, and/or Fluorescence in situ Hybridization (FISH) analysis; tissue or cells for analysis can be obtained at enucleation, resection, or by fine needle aspirate (FNA).
* Patients must have undergone adequate primary therapy; this can include enucleation, brachytherapy, proton beam radiotherapy, stereotactic irradiation, trans-scleral local resection, transretinal resection or diode laser thermotherapy
* Patients must have had chest X-ray and hepatic ultrasound or other imaging methods such as CT or MRI to eliminate distant disease
* Patients must have a performance status (ECOG) of < 2
* Patients must be entered within 56 days of completing primary therapy
* White blood count (WBC) ≥ 3.0 x 10^9/L
* Neutrophils ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* international normalized ratio (INR) and partial thromboplastin time (PTT) < 1.5 x upper limit of normal
* Hemoglobin ≥ 10 gm/100 ml
* Creatinine ≤ 2 mg/dl
* Bilirubin (total) ≤ 1.5 mg/dl
* Alanine transaminase (ALT) ≤ 1.5 x upper limit of normal
* Alkaline phosphatase ≤ 1.5 x upper limit of normal
* Aspartate aminotransferase (AST) ≤ 1.5 x upper limit of normal
* Patients must not have received any other systemic therapy for melanoma
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* All patients must be informed of the investigational nature of this study and must provide written informed consent in accordance with institutional and federal guidelines; a copy of the informed consent document signed by the patient must be given to the patient

Exclusion

* Patients with metastasis
* Patients that are pregnant or breastfeeding
* Patients may not be receiving any other investigational agents
* Patients with a history of immunodeficiency or autoimmune diseases are not eligible; patients requiring therapy with corticosteroids or other immunosuppressives are not eligible; patients requiring ongoing replacement therapy with physiologic doses of corticosteroids will be eligible.
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements are not eligible
* Patients who are known to be positive for HIV or Hepatitis B Surface Antigen (HepBAg)
* No patient may have had a malignancy other than a malignant melanoma, with the following exceptions: basal or squamous cell carcinomas of the skin; carcinoma in-situ of the uterine cervix; any malignancy treated with curative intent and in complete remission for > 3 years
* Patients with organ allografts

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-11-11 (Actual); Primary Completion 2015-07-25 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yogen Saunthararajah, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Binkley E, Triozzi PL, Rybicki L, Achberger S, Aldrich W, Singh A. A prospective trial of adjuvant therapy for high-risk uveal melanoma: assessing 5-year survival outcomes. Br J Ophthalmol. 2020 Apr;104(4):524-528. doi: 10.1136/bjophthalmol-2019-314461. Epub 2019 Aug 1. PMID 31371315

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Dacarbazine + Recombinant Interferon Alfa-2b: Patients receive dacarbazine IV on days 1 and 29. Beginning 4 weeks after the second dose of dacarbazine, patients receive recombinant interferon alfa-2b subcutaneously 3 times a week for 24 weeks in the absence of disease progression or unacceptable toxicity.
  recombinant interferon alfa-2b: Given subcutaneously (SC) 3 times a week for 24 weeks
  dacarbazine: Given IV on days 1 and 29
  laboratory biomarker analysis: Correlative studies obtained prior to therapy, every 8 weeks while on therapy, and then every 6 months during follow-up
Period: Overall Study
Arm/Group | Arm I: Dacarbazine + Recombinant Interferon Alfa-2b
Started | 38
Completed | 35
Not Completed | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All patients enrolled in study, regardless of treatment
Groups:
- Arm I: Dacarbazine + Recombinant Interferon Alfa-2b: Patients receive dacarbazine IV on days 1 and 29. Beginning 4 weeks after the second dose of dacarbazine, patients receive recombinant interferon alfa-2b subcutaneously 3 times a week for 24 weeks in the absence of disease progression or unacceptable toxicity.
  recombinant interferon alfa-2b: Given SC 3 times a week for 24 weeks
  dacarbazine: Given IV on days 1 and 29
  laboratory biomarker analysis: Correlative studies obtained prior to therapy, every 8 weeks while on therapy, and then every 6 months during follow-up
Arm/Group | Arm I: Dacarbazine + Recombinant Interferon Alfa-2b
Number analyzed (Participants) | 38
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 2
  30-39 years | 2
  40-49 years | 3
  50-59 years | 16
  60-69 years | 9
  70-79 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Disease-free Survival (DFS)
Description: DFS will be calculated from the date treatment starts to the date of documented recurrence or death. It will be summarized using the method of Kaplan and Meier. Treatment will be considered relatively ineffective in this population if the underlying 2-year DFS is <60%, whereas the combination will be considered promising if the underlying rate is >80%.
Time Frame: 5 years from time-of-enrollment
Population: All patients enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Dacarbazine + Recombinant Interferon Alfa-2b
Number analyzed (Participants) | 38
Participants | 8

2. Secondary Outcome: Number of Participants With Toxicity or Grade 4 Adverse Events Via CTCAE Version 3.0
Description: Number of participants with toxicity as defined as an underlying risk of >33% Grade 3 (non blood/bone marrow) or Grade 4 adverse events that are related to therapy, assessed by NCI CTCAE version 3.0
Time Frame: up to 32 weeks from start of study
Population: All patients enrolled on study regardless of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Dacarbazine + Recombinant Interferon Alfa-2b
Number analyzed (Participants) | 38
Participants | 2

3. Secondary Outcome: Changes in Plasma Biomarkers and Their Association With DFS
Description: Plasma levels of these markers will be summarized at baseline and over time quantitatively and graphically. Specific regulators of immune escape and tumor cell invasion identified in uveal melanoma gene array studies will be measured. Peripheral blood cells and plasma will be analyzed for granulysin (a measure of natural killer cells (NK) activity), beta2-microglobulin, autotoxin, lysophosphatidic acid (a product of autotaxin), matrix metalloproteinase-7, tissue inhibitor of matrix metalloproteinase, and soluble E-cadherin.
Time Frame: 5 yrs from start of treatment
Population: Information not collected
Arm/Group | Arm I: Dacarbazine + Recombinant Interferon Alfa-2b
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: During treatment up to 32 weeks
Arm/Group | Arm I: Dacarbazine + Recombinant Interferon Alfa-2b
All-Cause Mortality (participants affected / at risk) | 10/38
Serious Adverse Events (participants affected / at risk) | 2/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Dacarbazine + Recombinant Interferon Alfa-2b (N=38)
Constitutional Symptoms - Other (General disorders) | 1 (1)
Coagulation - Other (Blood and lymphatic system disorders) | 1 (1) — Pulmonary emboli to pulmonary arterial branches
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Dacarbazine + Recombinant Interferon Alfa-2b (N=38)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Lymphocele (Blood and lymphatic system disorders) | 2 (2)
Mood alteration - Anxiety (Nervous system disorders) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Ocular/Visual - vision impaired (Eye disorders) | 2 (2)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 2 (2)
Pain - Back (General disorders) | 2 (3)
Pain - Extremity-limb (General disorders) | 2 (2)
Pain - Joint (General disorders) | 2 (2)
Sweating (diaphoresis) (General disorders) | 2 (2)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (4)
Flushing (Skin and subcutaneous tissue disorders) | 3 (3)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3 (3)
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (5)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 3 (3)
Insomnia (General disorders) | 3 (4)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3)
Vision-flashing lights/floaters (Eye disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 4 (5)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 4 (7)
Vomiting (Gastrointestinal disorders) | 4 (4)
Allergic reaction/hypersensitivity (Immune system disorders) | 5 (5)
Anorexia (Gastrointestinal disorders) | 5 (5)
Pain - Muscle (General disorders) | 5 (5)
Pain - Generalized (General disorders) | 5 (5)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5 (5)
Mood alteration - Depression (Nervous system disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 7 (9)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 7 (12)
Pain - Head/headache (General disorders) | 8 (12)
Diarrhea (Gastrointestinal disorders) | 9 (10)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 10 (13)
Rigors/chills (General disorders) | 10 (15)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 12 (16)
Lymphopenia (Blood and lymphatic system disorders) | 12 (26)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 16 (21)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 17 (37)
Platelets (Blood and lymphatic system disorders) | 17 (23)
Nausea (Gastrointestinal disorders) | 24 (35)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 34 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes